CLINICAL TRIAL: NCT01640522
Title: Phase III Randomized Controlled Trial of a Collaborative Care Intervention to Manage Cancer Related Symptoms in Patients Diagnosed With Hepatobiliary Carcinoma
Brief Title: Comprehensive Electronic Cancer Support System for the Treatment of Cancer Related Symptoms
Acronym: CaSSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Steel, Director, Center for Excellence in Behavioral Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO07050143; K07CA118576 (NIH)
Record Dates: First submitted 2010-09-16; First posted 2012-07-13 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma; Primary Liver Cancer; Bile Duct Cancer; Pancreatic Cancer; Gallbladder Cancer; Colorectal Carcinoma; Liver Metastases
Keywords: Hepatocellular carcinoma; Cholangio carcinoma; Primary Liver Cancer; Bile Duct CancerPancreatic Cancer; Gallbladder Cancer; Colorectal Carcinoma; Other Primary Cancers with Liver Metastases
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bile Duct Neoplasms; Pancreatic Neoplasms; Gallbladder Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention versus standard of care
Who Masked: Outcomes Assessor
Masking Description: Only person evaluating outcomes
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collaborative Care Intervention (Experimental): Care coordinator facilitates the assessment and treatment of cancer-related symptoms
  Interventions: Other: Collaborative Care
- Enhanced Usual Care (Active Comparator): Upon evaluation of symptoms the patient will be referred for further assessment or treatment if indicated
  Interventions: Other: Enhanced usual Care

INTERVENTIONS:
Other: Collaborative Care — Collaborative care intervention to manage cancer-related symptoms
  Arms: Collaborative Care Intervention
Other: Enhanced usual Care
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of this study is to test the efficacy of a collaborative care intervention to manage cancer-related symptoms and improve health related quality of life in patients diagnosed with hepatobiliary carcinoma.

DETAILED DESCRIPTION:
The study is a collaborative care intervention designed to reduce pain, fatigue, and depressive symptoms and improve overall health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* biopsy, radiological, and/or biological evidence of hepatobiliary carcinoma
* age 18 years or older
* fluency in English. Exclusion criteria included:

Exclusion Criteria:

* current suicidal or homicidal ideation
* current psychosis or thought disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Depression | Change from baseline at 6 and 12 months
  Center for Epidemiological Studies-Depression scale

SECONDARY OUTCOMES:
Fatigue | Change from baseline at 6 and 12 months
  Functional Assessment of Cancer Therapy-Fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Steel, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States